CLINICAL TRIAL: NCT06602219
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose Ranging Study of LY4100511 (DC-853) for the Treatment of Adult Participants With Moderate-to Severe Plaque Psoriasis
Brief Title: A Study of LY4100511 (DC-853) in Adult Participants With Moderate-to-Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18845; J5C-MC-FOAB (Other: DCE853201)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY4100511 Dose 1 (Experimental): Participants will receive LY4100511 orally.
  Interventions: Drug: LY4100511
- LY4100511 Dose 2 (Experimental): Participants will receive LY4100511 orally.
  Interventions: Drug: LY4100511
- LY4100511 Dose 3 (Experimental): Participants will receive LY4100511 orally.
  Interventions: Drug: LY4100511
- Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4100511 — Administered orally
  Arms: LY4100511 Dose 1; LY4100511 Dose 2; LY4100511 Dose 3
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the safety and efficacy of LY4100511 in adult participants with moderate-to-severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of plaque psoriasis for 6 months before the baseline day 1 randomization
* Must have a body mass index (BMI) of 18 to 40 kilogram/square meter (kg/m2) (inclusive).
* Must be willing to discontinue topical and/or systemic therapies for psoriasis before the first dose of study intervention.
* Must agree to avoid prolonged exposure to the sun and to refrain from the use of tanning booths, sun lamps, and other sources of ultraviolet light during the study

Exclusion Criteria:

* Have had a clinically significant flare of psoriasis during the 12 weeks before the baseline, as assessed by the investigator.
* Have a history of erythrodermic psoriasis, generalized or localized pustular psoriasis, predominantly guttate psoriasis, or medication-induced or medication-exacerbated psoriasis.
* Have any known or suspected diagnosis of inflammatory conditions other than psoriasis and psoriatic arthritis, including but not limited to rheumatoid arthritis, sarcoidosis, IBD (Crohn's disease or ulcerative colitis), or systemic lupus erythematosus.
* Have a diagnosis of psoriatic arthritis requiring, or are currently receiving, systemic immunosuppressant medical treatment (including corticosteroids, immunosuppressants, and biologics).
* Have a current or recent acute, active infection. Participant must have no symptoms or signs of confirmed or suspected infection and must have completed any appropriate anti-infective treatment for at least 30 days before screening and up to randomization/baseline.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 75 | Week 12

SECONDARY OUTCOMES:
Percentage of Participants Achieving an sPGA Score of 0 (clear) or 1 (almost clear) with ≥2 grade Improvement from Baseline | Week 12
Percentage of Participants Achieving ≥50% Reduction in PASI score (PASI 50) | Week 12
Percentage of Participants Achieving ≥75% Reduction in PASI score (PASI 75) | Week 12
Percentage of Participants Achieving ≥90% Reduction in PASI score (PASI 90) | Week 12
Percentage of Participants Achieving 100% Reduction in PASI score (PASI 100) | Week 12
Percentage of Participants Achieving an sPGA Score of 0 or 1 | Week 12
Mean Change from Baseline in PASI Score | Week 12
Percent Change from Baseline in PASI Score | Week 12
Mean Change from Baseline in the Percentage of BSA Affected | Week 12
Percent Change from Baseline in the Percentage of BSA affected | Week 12
Pharmacokinetics (PK): Steady State Maximum Concentration of LY4100511 (Cmax,ss) | Predose up to 84 Days
PK: Steady State Trough Concentration (Ctrough,ss) | Predose up to 84 Days
Number of participants with one or more Adverse Event (s) (AEs), and Serious Adverse Event(s) (SAEs) considered by the by the investigator to be related to study drug administration | Baseline to Week 12
  A summary of AEs, SAEs and other non- serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events Module.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (58):
- United States (15):
  - Cahaba Dermatology Skin Health Center, Birmingham, Alabama
  - Dermatology Trial Associates, Bryant, Arkansas
  - Zenith Research, Inc., Beverly Hills, California
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Clinical Science Institute, Santa Monica, California
  - Driven Research, Coral Gables, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Renstar Medical Research, Ocala, Florida
  - GCP Global Clinical Professionals, LLC, St. Petersburg, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Endeavor Clinical Trials Center - Dermatology - Skokie, Skokie, Illinois
  - Lawrence J Green, M.D, LLC, Rockville, Maryland
  - Center for Clinical Studies, LTD.LLP, Webster, Texas
- Canada (8):
  - Interior Dermatology Centre - Probity - PPDS, Kelowna, British Columbia
  - Skin Care West, Nanaimo, British Columbia
  - Simcoderm Medical & Surgical Dermatology Centre, Barrie, Ontario
  - Dermatrials Research Inc., Hamilton, Ontario
  - Lovegrove Dermatology - Probity - PPDS, London, Ontario
  - DermEffects - Probity - PPDS, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
- Czechia (5):
  - Clintrial s.r.o., Prague, Praha 10
  - Pratia Pardubice a.s. - PRATIA - PPDS, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Pratia Prague s.r.o. - PRATIA - PPDS, Prague
  - Kozni ambulance Fialova, s.r.o. - CRC - PPDS, Prague
- Germany (6):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Praxis Dr. med. Virgil-Oreste Mihaescu Facharzt fr Dermatologie und STD, Augsburg, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus an der TU, Dresden
  - MensingDerma Research GmbH, Hamburg
- Hungary (4):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
  - Allergo-Derm Bakos Kft, Szolnok, Jász-Nagykun-Szolnok
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - MedMare Bt, Veszprém
- Japan (9):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Medical Corporation Kojinkai Sapporo Skin Clinic, Sapporo, Hakkaido
  - Katahira Dermatology Urology Clinic, Kagoshima, Kagoshima-ken
  - Ohyama Dermatology Clinic, Kumamoto, Kumamoto
  - Kume Clinic, Sakai-shi, Osaka
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Tachikawa Dermatology Clinic, Tachikawa, Tokyo
  - Shirasaki dermatology clinic, Takaoka, Toyama
  - Igarashi Dermatological Clinic, Tokyo
- Poland (11):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Cityclinic Przychodnia Lekarsko Psychologiczna Matusiak Spółka Partnerska, Wroclaw, Lower Silesian Voivodeship
  - Clinical Best Solutions, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Fryderyka Chopina w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk, Pomeranian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa, Silesian Voivodeship
  - Laser Clinic Dermatologia Laserowa Medycyna Estetyczna, Szczecin, West Pomeranian Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice
  - Centrum Medyczne Reuma Park NZOZ, Warsaw
  - Dermoklinika Centrum Medyczne s.c. M. Kierstan J. Narbutt A. Lesiak, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/